CLINICAL TRIAL: NCT06824805
Title: Hypertension, Ethnicity and Exercise Trial
Acronym: HYPE2X
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Véronique Cornelissen, Professor, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 183/2020
Record Dates: First submitted 2025-02-10; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- isometric handgrip exercise (Active Comparator): 4x2 minutes of isometric handgrip exercise
  Interventions: Behavioral: Exercise
- control (No Intervention): seated control session
- Aerobic exercise (Experimental): aerobic exercise at 40-60% HRres
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — aerobic exercise for 30 minutes at 40-60% HRres
  Arms: Aerobic exercise; isometric handgrip exercise

SUMMARY:
The main aim of this study is to investigate the acute effects of a single bout of isometric handgrip exercise (IHG) and a single bout of aerobic endurance exercise (AEX) on blood pressure, both immediately after exercise and during the subsequent activities of daily living in patients with high-normal to grade 1 hypertension of South-Asian or African descent living in Suriname.

ELIGIBILITY:
Inclusion Criteria:

* • Age 18 - 65 years

  * Patients with high- normal BP (SBP: 130 - 139 mmHg or and DBP: 85 - 89 mmHg) or stage I hypertension (SBP: 140 - 159 mmHg or DBP: 90 - 99 mmHg) according to the ESC/ESH guidelines [15]
  * Asian or African descent
  * Do not meet the level of physical activity recommended by the WHO based on self-report [15]
  * Non-medicated patients or patients using a maximum of 2 antihypertensive drugs

Exclusion Criteria:

* • Functional or mental limitation limiting the correct execution of an exercise bout

  * History of ischemic stroke, autonomic neuropathy, cardiovascular, renal, or pulmonary disease by self-report
  * Diabetes type I or II
  * Pregnancy
  * The presence of exercise induced signs of myocardial ischemia or complex ventricular arrhythmia during CPET
  * Patients using three or more antihypertensive drugs or patients with resistant hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
office blood pressure at 30 minutes post exercise | 30 minutes postexercsie
  office blood pressure at 30 minutes post exercise

SECONDARY OUTCOMES:
daytime blood pressure | mean of 8 hours after the intervention
  daytime ambulatory blood pressure (8 hours after the intervention)

CONTACTS AND LOCATIONS:
Locations (1):
- Anton De Kom University, Paramaribo, Suriname

IPD SHARING:
Plan to Share IPD: Undecided